CLINICAL TRIAL: NCT05633706
Title: Evaluation of the Small Intestine Microbiome Aspiration (SIMBA) Capsule for Small Intestinal Dysbiosis
Brief Title: Evaluation of the SIMBA Capsule for Small Intestinal Dysbiosis
Status: Recruiting | Type: Observational
Sponsor: Nimble Science Ltd. (Industry)
Collaborators: Mitacs (Industry); University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CTC-22-0096
Record Dates: First submitted 2022-09-26; First posted 2022-12-01 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Irritable Bowel Syndrome; Crohn Disease; Celiac Disease; Ulcerative Colitis; Functional Dyspepsia; Type 2 Diabetes; Healthy
Keywords: Microbiome
MeSH Terms: conditions — Irritable Bowel Syndrome; Crohn Disease; Celiac Disease; Colitis, Ulcerative; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fluid from the small intestine, stool, saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Healthy: Not belonging to the other cohorts as described below.
  Interventions: Device: fluid biopsy capsule
- Irritable Bowel Syndrome: As confirmed by diagnosis and/or PI assessment, and measured via patient response to validated questionnaires - no interventions applied.
  Interventions: Device: fluid biopsy capsule
- Crohns Disease: As confirmed by diagnosis and/or PI assessment, and measured via patient response to validated questionnaires - no interventions applied.
  Interventions: Device: fluid biopsy capsule
- Ulcerative Colitis: As confirmed by diagnosis and/or PI assessment, and measured via patient response to validated questionnaires - no interventions applied.
  Interventions: Device: fluid biopsy capsule
- Celiac Disease: As confirmed by diagnosis and/or PI assessment, and measured via patient response to validated questionnaires - no interventions applied.
  Interventions: Device: fluid biopsy capsule
- Functional Dyspepsia: As confirmed by diagnosis and/or PI assessment, and measured via patient response to validated questionnaires - no interventions applied.
  Interventions: Device: fluid biopsy capsule
- Type 2 Diabetes: As confirmed by diagnosis and/or PI assessment, and measured via patient response to validated questionnaires - no interventions applied.
  Interventions: Device: fluid biopsy capsule

INTERVENTIONS:
Device: fluid biopsy capsule — Collection of a fluid biopsy from the small intestine via ingestible capsule

SUMMARY:
The SIMBA Capsule is a small, single-use, ingestible capsule that allows for the non-invasive sampling of small bowel contents using purely mechanical means. The study will compare the microbial and metabolomics analysis from the sample collected with the capsule series, to same-participant symptom questionnaires and stool microbial analysis.

DETAILED DESCRIPTION:
The investigators primary goal is to assess the correlation of gut symptoms from various disease states with the dysbiosis of the small intestinal microbiome and metabolites collected by the SIMBA capsule, and as identified and measured by metagenomic sequencing and/or metabolomics approaches. The process consists of ingestion and collection of up to 4 SIMBA capsules, on up to 2 separate occasions, along with collection of a stool sample at the same time. Participants will also fill out a series of questionnaires on medical history and lifestyle inputs (eg. diet, exercise, mental health) GI symptoms, anxiety, and depression. The investigators ultimate goal will be to develop a better understanding of how the small intestinal microbiome might play a role in symptom generation, to establish whether the SIMBA capsule can find a signature of dysbiosis which can be used as a biomarker for a number of functional gut disorders.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Aged between 18 and 80 years.
2. No previous diagnosis of Celiac Disease, Ulcerative Colitis, Crohn's disease, IBS, Functional Dyspepsia, and T2D by participant self-report (Control group).
3. Prior diagnosis of Celiac Disease, Ulcerative Colitis, Crohn's disease, IBS, or Functional Dyspepsia, and T2D by a relevant physician, nutritionist, naturopath, etc, and willingness to provide documentation to confirm this diagnosis or have a consultation with the PI. (Disease group).
4. Ability to understand and provide informed consent.
5. Ability and willingness to meet the required schedule, study interventions, and questionnaire requirements.
6. No planned change in diet or medical interventions during the study duration.

Exclusion Criteria

1. Known disease which, in the investigator's opinion, would lead to intestinal structuring or obstruction with a risk of capsule non-excretion (particular diseases which would be assessed on a case-by-case basis would include, achalasia, eosinophilic esophagitis, cancer diagnosis or treatment within the past year, or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months prior to enrollment are acceptable). The main deciding factor would be a history of obstructive symptoms in the previous 3 months prior to entry.
2. Use of any medications or having undergone procedures in the previous week that could substantially alter gastrointestinal motor function (e.g., opioids, anticholinergics, laxatives, or GLP-1 analogues).

   1. Stimulant laxative use (includes bisacodyl/Dulcolax, senna/Senekot, cascara, or fibre supplments) is allowed if it is kept unchanged in the week prior to the SIMBA Capsule ingestion. Osmotic laxatives (polyethylene glycol (PEG; other trade names), milk of magnesia, lactulose), stool softeners (docusate; other trade names) or secretagogues (linaclotide/Constella, plecanatide/Trulance, tenapanor/Ibsrela should not be used within 7 days of taking the SIMBA capsules.
   2. Prokinetics use is allowed if kept unchanged in the week prior to the SIMBA Capsule ingestion (includes domperidone, metoclopramide, prucalopride). Inconsistent use of prokinetics will be evaluated by the PI.
   3. PPI or H2RA use. Must be able to discontinue PPI or H2RA medications 48hrs prior to SIMBA capsule ingestion, medication can be resumed 4 hours after ingestion.
3. History of oropharyngeal dysphagia or other swallowing disorder with a risk of aspiration of the capsule.
4. History of known structural gastrointestinal abnormalities such as strictures or fistulas leading to mechanical obstruction
5. History of abdominal radiation treatment
6. Females of childbearing age who are pregnant or lactating by self-report. (should an X-ray be required for confirmation of capsule passage, a urine pregnancy test will be administered beforehand).
7. No antibiotics, or colon cleanses/bowel prep for 2 weeks.
8. < 2 bowel movements per week (Control Group only).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 300 individuals, females or males will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of bacterial composition with gastrointestinal disease states as assessed by PLS-DA mapping. | baseline, pre-procedure
  The bacterial composition of healthy control fluid biopsy is compared to the bacterial composition of participants with diagnosed gastrointestinal diseases, to aid in gastrointestinal disease biomarker discovery.

SECONDARY OUTCOMES:
Correlation of bacterial composition with dietary intake as assessed by PLS-DA mapping. | baseline, pre-procedure
  Fluid biopsy bacterial composition correlated with self-reported long-term and short-term preferred variations in intake of dietary fiber and organic food.

OTHER OUTCOMES:
Usability of SIMBA capsule in various disease states as assessed by SIMBA-experience questionnaires. | immediately after the procedure
  Participant feedback on SIMBA capsule usage experience will inform usability data.
Comparison of SIMBA fluid biopsy microbial composition to stool microbial composition as assessed by 16s rRNA metagenomic analysis. | baseline, pre-procedure
Correlations of bacterial composition with anxiety (GAD-7) scores as assessed by PCoA mapping, alpha and beta diversity analysis. | baseline, pre-procedure
Correlations of bacterial composition with depression (PHQ-8) scores as assessed by PCoA mapping, alpha and beta diversity analysis. | baseline, pre-procedure
Correlations of bacterial composition with self-reported lifestyle behaviours as assessed by PCoA mapping, alpha and beta diversity analysis. | baseline, pre-procedure
Number of participants with device-related adverse events as assessed by an independent Data Safety Monitoring Board. | through study completion, an average of 8 days
Evaluate the usability of excreted SIMBA Capsule retrieval procedures as assessed by retrieval-experience questionnaire feedback. | immediately after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Chris Andrews, MD, Principal Investigator — Nimble Science Ltd.; Matthew Woo, MD, Principal Investigator — Nimble Science Ltd.
Locations (1):
- Nimble Science, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No